CLINICAL TRIAL: NCT02278458
Title: Phase I, Open-label, Dose-escalation Study to Evaluate the Safety and Tolerability of Icotinib Combined With Gemcitabine as First-line Treatment in Locally Advanced, Unresectable or Metastatic Pancreatic Cancer
Brief Title: Combination of Icotinib and Gemcitabine as First-line Treatment in Pancreatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV70
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — icotinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- icotinib plus gemcitabine (Experimental): Three dose of icotinib are designed to be evaluated, 125 mg three times per day, 250 mg three times per day, and 375 mg three times per day. Dose escalations are based on predefined dose escalation decision rules. The Maximum Administered Dose (MAD) was reached at the dose level when at least 30% patients developed a dose limited toxicity.
  Gemcitabine: 1000 mg/m2 on Days 1, 8, and 15 of a 28 day cycle by IV administration every 4 weeks.
  Interventions: Drug: icotinib; Drug: Gemcitabine

INTERVENTIONS:
Drug: icotinib — Three dose levels of icotinib are designed to be evaluated, 125 mg three times per day, 250 mg three times per day, and 375 mg three times per day. Dose escalations are based on predefined dose escalation decision rules. The Maximum Administered Dose (MAD) was reached at the dose level when at least 30% patients developed a dose limited toxicity.
  Other Names: Commana
Drug: Gemcitabine — Gemcitabine: 1000 mg/m2 on Days 1, 8, and 15 of a 28 day cycle by IV administration every 4 weeks.
  Other Names: Gemzar

SUMMARY:
Research Hypothesis: icotinib administered in combination with gemcitabine has an acceptable safety profile in subjects with locally advanced, unresectable or metastatic pancreatic adenocarcinoma.The primary objective is to determine the safety profile of icotinib in combination with gemcitabine in subjects with locally advanced, unresectable or metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, unresectable or metastatic pancreatic cancer by histologic or cytologic confirmation without previous chemotherapy or target therapy.
* ECOG Performance Status of 0 to 1.
* Adequate organ function as defined by study-specified laboratory tests.
* Signed informed consent form.
* Willing and able to comply with study procedures.

Exclusion Criteria:

* Previous chemotherapy or target therapy.
* Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, immune or other medical conditions.
* Systemically active steroids.
* Another investigational product within 28 days prior to receiving study drug.
* Major surgery or significant traumatic injury (or unhealed surgical wounds) occurring within 28 days prior to receiving study drug.
* Infection with HIV, hepatitis B or C at screening.
* Pregnant or lactating.
* Conditions, including alcohol or drug dependence, or intercurrent illness that would affect the patient's ability to comply with study visits and procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-01 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The number of patients who suffer adverse events | 24 months

SECONDARY OUTCOMES:
Tumor response assessed by RECIST 1.1 | 3 months
Progression-free survival | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiao Zhang, MD, Principal Investigator — Cancer Hospital of Harbin Medical University
Locations (3):
- China (3):
  - Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Bethune First Hospital of Jilin University, Changchun, Jilin
  - First Affiliated Hospital of China Medical University, Shenyang, Liaoning